CLINICAL TRIAL: NCT04072523
Title: An Observational, Cross Sectional Study to Assess the Prevalence of Heart Failure in Type 2 Diabetes Patients in India
Brief Title: An Observational Study to Assess the Prevalence of Heart Failure in Type 2 Diabetes Patients
Acronym: HF-Registry
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00300
Record Dates: First submitted 2019-08-27; First posted 2019-08-28 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes, Heart Failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Study Investigational Product NA: Patients : Type 2 Diabetic Patients

SUMMARY:
An Observational Study to assess the Prevalence of Heart Failure in Type 2 Diabetes Patients in India.

DETAILED DESCRIPTION:
This is a cross sectional, observational, multi-centre study to be conducted at 40 centres in India. The study targets to enrol 1000 patients with approx. 25 patients per site. The study would enrol Type 2 Diabetes Mellitus patients who provide written informed consent. No study medication will be prescribed or administered as a part of study procedure. Patients, who have been treated as per Investigators' routine clinical practice will be screened for enrolment in study. The study will be initiated after obtaining written approval of Independent Ethics Committee (IEC) /Institutional Review Board (IRB).

ELIGIBILITY:
Inclusion Criteria:

* Both men and women aged ≥ 18 years
* Diagnosed with type 2 diabetes (as per ADA Criteria)
* Duration of diabetes for 1 year or more
* Willing to provide the informed consent

Exclusion Criteria:

* Patients with evidence of coronary artery disease - CAD (based on the clinical expertise of the physician).
* Patients who were previously diagnosed with heart failure.
* Patients with evidence of valvular disease based on clinical judgement of the Principle Investigator (PI).
* Current treatment with digoxin.
* History of symptoms of peripheral artery disease, chronic obstructive pulmonary disease and arrhythmias.
* Patients diagnosed with stage III/IV CKD
* Diabetes other than type 2 diabetes mellitus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: type 2 diabetes mellitus patients
Sampling Method: Non-Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Left Ventricular dysfunction | 1 day
  based on the BNP levels and echocardiography results.

SECONDARY OUTCOMES:
Correlation of Left ventricular dysfunction and heart failure | 1 day
  With demographics and comorbidities of the patients to assess relation between them.

CONTACTS AND LOCATIONS:
Locations (16):
- India (16):
  - Research Site, Ahemdabad, Gujarat
  - Research Site, Rajkot, Gujarat
  - Research Site, Rohtak, Haryana
  - Research Site, Bangalore, Karnataka
  - Research Site, Kochi, Kerala
  - Research Site, Mumbai, Maharashtra
  - Research Site, Delhi, New Delhi
  - Research Site, Amritsar, Punjab
  - Research Site, Chandigarh, Punjab
  - Research Site, Jalandhar, Punjab
  - Research Site, Ludhiana, Punjab
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Hyderabad, Telangana
  - Research Site, Kanpur, Uttar Pradesh
  - Research Site, Kolkata, West Bengal
  - Research Site, Delhi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00300&attachmentIdentifier=131457da-2eba-4d49-949a-00655d77daf5&fileName=Redacted_Study_Report_Synopsis_V1.0_D1843R00300.pdf&versionIdentifier=